CLINICAL TRIAL: NCT07092098
Title: The Effects of Transcranial Direct Current Stimulation Combined With Resistance Training on Motor Learning in Healthy Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TEOTDCSCWRTOMLIHYA
Record Dates: First submitted 2025-07-20; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Resistance Training; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tDCS combined with resistance training (Experimental)
  Interventions: Combination Product: tDCS combined with resistance training
- Resistance training alone (Experimental)
  Interventions: Behavioral: Resistance training
- tDCS alone (Experimental)
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator)
  Interventions: Device: sham tDCS

INTERVENTIONS:
Combination Product: tDCS combined with resistance training — Transcranial direct current stimulation combined with resistance training
  Arms: tDCS combined with resistance training
Behavioral: Resistance training — low-limb resistance training
  Arms: Resistance training alone
Device: tDCS — Transcranial direct current stimulation
  Arms: tDCS alone
Device: sham tDCS — Sham transcranial direct current stimulation
  Arms: Sham tDCS

SUMMARY:
This study aimed to investigate whether six weeks of tDCS combined with lower-limb resistance training could enhance motor learning in healthy young adults and examined the persistence of any observed benefits.

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected-to-normal vision
* right-handed

Exclusion Criteria:

* color blindness
* color weakness
* dyslexia
* history of smoking
* cardiovascular diseases
* personal or family history of mental illness

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Sequence Reaction Time Task | Motor learning was assessed at before intervention, after three and six weeks of intervention, and one week post-intervention.
  In this task, a white circle appears above one of four horizontally arranged white squares on the computer screen with black background. Participans were instructed to press the proper button on the response pad (buttons H, J, K, L) using the corresponding finger of the right hand (index finger for button H, middle finger for button J, ring finger for button K, and small finger for button L) when the white circle appeared at the left side, middle-left side, middle-right side, or right side of the computer screen, respectively. Each session consists of eight blocks, with each block comprising 120 trials.